CLINICAL TRIAL: NCT01885026
Title: Substance-use Focused Screening and Brief Intervention as a Complement to Internet-based Psychiatric Treatment for Depression, Panic Disorder or Social Phobia: A Randomized Controlled Trial
Brief Title: Substance-focused SBI as a Complement to Internet-based Psychiatric Treatment: RCT
Acronym: eScreeniPsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/1138-31/1; KI 4-2007/2013 (Other: Karolinska Institutet, Legal Dept)
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Substance Use Disorders (SUD)
Keywords: Randomized Controlled Trial; Alcohol; Drugs; Internet; Screening; Brief intervention
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- eScreen (Experimental): Web based self-monitoring of problematic alcohol and drug use, and Internet-based treatment for depression or anxiety
  Interventions: Behavioral: eScreen; Behavioral: Internet-based treatment for depression or anxiety
- Control (Experimental): Assessment only of alcohol and drug use and Internet-based treatment for depression or anxiety
  Interventions: Behavioral: Assessment only of alcohol and drug use.; Behavioral: Internet-based treatment for depression or anxiety

INTERVENTIONS:
Behavioral: eScreen — Access to the eScreen platform offering assessment of alcohol and drug use, with automated feedback on problematic or non-problematic use. Follow-up over time based on user needs.
  Arms: eScreen
Behavioral: Assessment only of alcohol and drug use. — Assessment of alcohol and drug use at baseline and follow-up.
  Arms: Control
Behavioral: Internet-based treatment for depression or anxiety — Internet-based treatment for primary diagnoses of depression, panic anxiety or social phobia.

SUMMARY:
Objectives: This study evaluates the efficacy of eScreen for internet psychiatry patients treated for major depressive disorder, panic anxiety and social phobia. The eScreen brief Internet intervention for problematic alcohol and drug use offers self-screening, in-depth self-reporting, personalized feedback and treatment recommendations as well as an electronic diary. Progress over time is shown in diagrams detailing consumption levels.

Method: This is a two-armed randomized controlled design, measuring outcomes in terms of changes in problematic alcohol use up to one year after study recruitment. Participants with problematic alcohol use (AUDIT >7 for men and >5 for women) and/or problematic drug use (DUDIT > 1 for both men and women) are randomized into one of two groups: T1, eScreen referral or Control group. Outcomes on alcohol and drug use as well as health-related symptoms are assessed after 3, 6 and 12 months.

The hypothesis is that the group receiving the eScreen intervention will reduce their alcohol/drug use to a larger extent than the control group at follow-up compared to the baseline level.

DETAILED DESCRIPTION:
This study evaluated the efficacy of eScreen for internet psychiatry patients treated for major depressive disorder, panic anxiety and social phobia. The eScreen brief Internet intervention for problematic alcohol and drug use offers self-screening, in-depth self-reporting, personalized feedback and treatment recommendations as well as an electronic diary. Progress over time is shown in diagrams detailing consumption levels. The design was a two-armed randomized controlled design, measuring outcomes in terms of changes in problematic alcohol use up to one year after study recruitment. Participants with problematic alcohol use (AUDIT >7 for men and >5 for women) and/or problematic drug use (DUDIT > 1 for both men and women) were randomized into one of two groups: T1, eScreen referral or Control group. Outcomes on alcohol and drug use as well as health-related symptoms are assessed after 3, 6 and 12 months.

The hypothesis was that the group receiving the eScreen intervention would reduce their alcohol/drug use to a larger extent than the control group at follow-up compared to the baseline level. The results have not yet been analyzed due to technical issues. However, qualitative interviews have been conducted with participants and our intention is to publish the qualitative results in tandem with the quantitative results available.

ELIGIBILITY:
Inclusion Criteria:

AUDIT >7 for men and AUDIT >5 for women, and/or DUDIT >0

Exclusion Criteria:

DUDIT = 0 and AUDIT <8 (men) or <6 (women)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the total AUDIT-C score | 3, 6 and 12 months
  The primary outcome measure for this trial is the change in the total AUDIT score for the first three AUDIT questions, as a measure of alcohol consumption only, referred to as the AUDIT-C.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | 3, 6 and 12 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems).

OTHER OUTCOMES:
Changes in health parameters over time | 3, 6 and 12 months
  Health-related questions on wellbeing, sleep, concentration, energy, social life, sadness and current life meaning, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Center for Psychiatric Research, Stockholm, Sweden

REFERENCES:
- [Background] Sinadinovic K, Berman AH, Hasson D, Wennberg P. Internet-based assessment and self-monitoring of problematic alcohol and drug use. Addict Behav. 2010 May;35(5):464-70. doi: 10.1016/j.addbeh.2009.12.021. Epub 2010 Jan 4. PMID 20092953
- [Background] Sinadinovic K, Wennberg P, Berman AH. Targeting problematic users of illicit drugs with Internet-based screening and brief intervention: a randomized controlled trial. Drug Alcohol Depend. 2012 Nov 1;126(1-2):42-50. doi: 10.1016/j.drugalcdep.2012.04.016. Epub 2012 May 20. PMID 22613182
- [Background] Sinadinovic K, Wennberg P, Berman AH. Internet-based screening and brief intervention for illicit drug users: a randomized controlled trial with 12-month follow-up. J Stud Alcohol Drugs. 2014 Mar;75(2):313-8. doi: 10.15288/jsad.2014.75.313. PMID 24650825
- See also: Link to participant registration site. — http://ipsy.epop.se